CLINICAL TRIAL: NCT04973956
Title: Influencia de la Ansiedad en el Aprendizaje Motor de Una Tarea Manual Precisa y en la Capacidad de Imaginación Motora
Brief Title: Influence of Anxiety on Motor Learning and Motor Imagery Ability in Young Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susana Nunez Nagy (Other)
Collaborators: University of Alcala (Other); Universidad Complutense de Madrid (Other); European University of Madrid (Other); Claude Bernard University (Other)
Responsible Party: Sponsor-Investigator, Susana Nunez Nagy, PhD. Associate Professor of Physiotherapy, University of Alcala
Organization: University of Alcala (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CEID2022/2/036_3
Record Dates: First submitted 2021-06-24; First posted 2021-07-22 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Anxiety
Keywords: Anxiety; Motor Learning; Memory; Motor Imagery Ability
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: As participants complete the State-Trait Anxiety Inventory, and are found to be anxiety, they will be randomised in parallel to one of the two intervention groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant does not know what the other participants are doing, the researcher knows which study and group the subject is in, but only sets up the computerized presentations for each group and assigns folders within the computer that collects the data, thus avoiding a possible information bias, and finally, another researcher blind to the intervention will analyse the data to obtain the results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation group (Active Comparator): This group will perform the APMR
  Interventions: Other: Relaxation
- Control group (Active Comparator): This group will perform the control intervention
  Interventions: Other: Control

INTERVENTIONS:
Other: Relaxation — This group will perform the APMR. This intervention consists of a standardized 20 min session in which subjects are asked to sequentially tense and relax various muscle groups. To do so, participants will listen to an audio with relaxation instructions while seated in a reclining seat and dimmed lighting.
  Arms: Relaxation group
Other: Control — No intervention
  Arms: Control group

SUMMARY:
In motor learning, to consider that movements are produced by the cooperation and combination of many brain structures and are influenced by the emotions to which individuals are subjected is essential. Several neural circuits have been identified that closely link the emotional system and the motion control system.

Anxiety is defined by persistent and excessive worries that do not disappear even in the absence of the stressor. Anxiety has been found to produce inefficiencies in information processing, which can result in performance deficits, as well as self-reported anxiety has been linked to poorer working retrieval performance. In these stress and anxiety contexts, relaxation techniques have been widely used to reduce psychophysiological arousal levels.

Understanding how movement, emotions and interactions are regulated is significant because of the large number of movements humans perform. Of these, manual tasks represent precise movements that require the integration of many elements by the nervous system to perform these tasks successfully. How anxiety influence the way manual tasks are learned is still unknown.

On the other hand, motor imagery (MI) is a cognitive process that is an important contributor to how movements are planned and executed. The use of MI has been recommended to improve movement learning and task execution. Knowing MI capacity is essential for creating effective and individualized MI programs. However, how a relax intervention can affect the motor imagery ability in anxiety people is still unknown.

The aim of our study was to find out whether a relaxation intervention prior to MI practice in subjects with anxiety can influence the learning of a precise manual task not previously trained on four parameters of fine motor control: time, error, speed, and accuracy. On the other hand, the aim is to determine if the ability of internal visual, external visual, and kinaesthetic imagery varies when the anxiety participants are subjected to relaxation.

The investigators expect that participants with anxiety, to whom relaxation is induced, will show better motor performance on the fine motor task and better motor imagery ability. In contrast, the investigators expect that participants with anxiety, to whom relaxation is not induced, will show poorer motor performance on the fine motor task and poorer motor imagery ability.

DETAILED DESCRIPTION:
In order to meet the study objectives of determining and quantifying the effects of relax in anxiety people on learning a precise manual task and on motor imagery ability, this study will be conducted. The development of the study will take place in a conditioned room belonging to the University of Alcalá, the Complutense University of Madrid, the European University of Madrid, or Claude Bernard University Lyon 1. The study may also be carried out in other Spanish and international university centers, subject to the consent and permission of the respective centres. The study will be carried out by all national and international laws, regulations, and recommendations.

The study design will be longitudinal, experimental, randomized, and double-blind, as specified in the present registry.

The study population will be composed of participants who are undergraduate and postgraduate students at the university centers where the study will be carried out, from which the participants will be recruited. All participants included in the study must meet the study selection criteria and participate voluntarily after reading the information sheet and signing the informed consent form.

The study will consist of two intervention groups, both groups will have anxiety measured with the State-Trait Anxiety Inventory (STAI) and then be randomized to either the relaxation intervention group or the control group. Each group will consist of a minimum number of 20 subjects to be able to study the desired effect.

After each participant freely chooses to participate in the study, an initial questionnaire will be administered to ensure that the participants meet the criteria for inclusion in the study. At this point, the participants will be coded by assigning them a number, which will serve to identify each participant throughout the study. Participants will take the STAI, one of the most widely used instruments for the self-reported assessment of anxiety. Participants with scores indicative of anxiety will be included in the study. Included participants will be randomized through sealed envelopes stratified by gender to one of two experimental groups: relaxation or control. They will also take the Edinburgh Handedness Inventory (EHI) to determine the participant's laterality, and the Movement Imagery Questionnaire-3 (MIQ-3) to measure internal visual, external visual, kinaesthetic imagery capacity. At the same time of MIQ-3, the experimenter will record the execution and imagery times were recorded (for subsequent calculation of the time discrepancy between executed and imagery as a measure of temporal congruence between them).

Depending on the group to which the participants have been assigned, the participants of the relaxation group will perform a relaxation intervention using the Abbreviated Progressive Muscle Relaxation technique (APMR). This intervention consists of a standardized 20 min session in which subjects are asked to sequentially tense and relax various muscle groups. To do so, participants will listen to an audio with relaxation instructions while seated in a reclining seat and dimmed lighting. Despite its brevity, this relaxation technique has been shown to be effective in reducing anxiety and has been shown to produce cognitive, behavioral, and physiological relaxation. On the other hand, participants in the control group did not receive a relaxation intervention. After the relaxation or control, participants will learn a precise manual task with the non-dominant hand. The task will consist of going over a 127 mm circumference on a graphics tablet at a rate of 2 seconds per lap, which will be set by a metronome using a wireless pen that will leave no trace of ink but will store the data in the MATLAB program via the graphics tablet. Thus, data from the acquisition process and short-term retrieval of the task will be recorded. Afterward, there will be a 20-minute break during which participants will perform the MIQ-3 and the experimenter will record the execution and imagery times again.

In addition, during all experiments, electrodermal activity and heart rate variability will be recorded using the Empatica E4 physiological variable measurement wristband. This measurement of physiological variables will serve to confirm a significant relax effect has been generated in the relaxation group.

The analysis and processing of data from MATLAB version R2020b, and the Empatica E4 wristband will be performed using Rstudio statistical software and Kubios HRV software (for HRV analysis).

First, appropriate statistical analyses will be performed to see if the data are distributed according to a standard curve and to assess the influence of sex and age.

Subsequently, the descriptive analysis of the relative and absolute frequencies for the qualitative variables of gender and age will be carried out, and their homogeneity will be tested using the Chi-square test. The descriptive analysis of the quantitative variables of time, error, speed, accuracy, electrodermal activity, heart rate variability, motor imagery capacity and discrepancy times also be carried out. If the variable conforms to the normal, the mean, range, and standard deviation shall be calculated. If the variables do not conform to the normal, non-parametric tests will be performed.

Comparative analysis will be performed using mixed ANOVA to see the differences in the mean values respective to motor control (time, error, speed, and accuracy). A further ANOVA analysis will take place for imagery ability (motor imagery capacity and discrepancy times), comparing the results obtained at the two respective points during the experiment.

The effect of learning between laps will be analyzed by repeated-measures ANOVA comparing each motor control measurement parameter with respect to the lapping factor. Electrodermal activity, and heart rate variability during the relaxation intervention will also be studied by repeated-measures ANOVA.

For hypothesis testing, a significance level of 0.05 will be set.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 35 years of age.
* Normal or corrected vision specifying the method of correction.
* Normal or corrected hearing specifying method of correction.
* Unfamiliar with the assessment and uses of motor imagery.
* Presence of State-Trait Anxiety Inventory scores corresponding to anxiety.

Exclusion Criteria:

* Subjects who have suffered fractures, dislocations, or traumatic processes in any segment of the non-dominant upper limb or fingers, wrist, or elbow of the dominant upper limb in the last 6 months.
* Subjects with learning disabilities or problems in reading or writing.
* Subjects with a history of any neurological disease, cardiovascular disease, myopathic disease, epileptic seizure, absence seizure, sleep apnoea, chronic fatigue syndrome, or fibromyalgia.
* Taking any medication to suppress anxiety, to sleep, antidepressants, antihistamines, muscle relaxants, psychotropic, or other medications that interfere with the nervous system.
* Intake of nervous system depressants or stimulants such as caffeine or theine in the last 8 hours.
* Presence of localised skin lesion or disease in the wrist area.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Trayectory error | During manual task performance in acquisition, short-term retrieval, and long-term retrieval
  It shall be the sum of the error between each of the points defining the path of the circumference. Pixels squared shall be considered as the unit of length measurement. To be recorded and measured with MATLAB. To be recorded and measured with MATLAB.
Timing error | During manual task performance in acquisition, short-term retrieval, and long-term retrieval
  It is the absolute value of the difference between the duration of 2 seconds requested from the subjects and the total time elapsed in the execution of the trajectory. It shall be expressed in seconds (s). It shall be recorded and measured using MATLAB.
Timing accuracy | During manual task performance in acquisition, short-term retrieval, and long-term retrieval
  The ability of the subject to learn the task at the requested rate of 2 seconds per lap. It shall be expressed in square pixels per second. It shall be recorded and measured by MATLAB.
Task accuracy | During manual task performance in acquisition, short-term retrieval, and long-term retrieval
  It shall be the ability of the subject to learn at any rate. It shall be expressed in pixels per second. It shall be recorded and measured by MATLAB.
Motor Imagery Capacity | Before induction of acute stress and in the resting period between short-term and long-term retrieval after induction of acute stress
  This will be measured using the Movement Imagery Questionnaire-3, differentiating between the kinaesthetic, external visual and internal visual imagination subscales, each scored on a Likert scale from 1 to 7.
Discrepancy time | Before induction of acute stress and in the resting period between short-term and long-term retrieval after induction of acute stress
  It will be the difference between the execution times and imagery of the MIQ-3 items. It will be measured with a stopwatch by the experimenter.

SECONDARY OUTCOMES:
Electrodermal Activity | During the procedure
  The skin conductance level shall be analyzed in terms of tonic Electrodermal Activity. It shall be recorded and measured by Empatica E4 wristband.
Heart Rate Variability | During the procedure
  It will be analysed in the frequency domain, in its low and high frequency bands and in the ratio between them. It shall be recorded and measured by Empatica E4 wristband.

CONTACTS AND LOCATIONS:
Overall Officials: Sara T Trapero Asenjo, Master, Principal Investigator — University of Alcala; Susana N Núñez Nagy, PhD, Study Director — University of Alcala; Sara F Fernández Guinea, PhD, Study Director — Universidad Complutense de Madrid
Locations (4):
- Claude Bernard University Lyon 1, Villeurbanne, Auvergne-Rhône-Alpes, France
- Spain (3):
  - University of Alcalá, Alcalá de Henares, Madrid
  - Complutense University of Madrid, Pozuelo de Alarcón, Madrid
  - European University of Madrid, Villaviciosa de Odón, Madrid

REFERENCES:
- [Background] Coombes SA, Cauraugh JH, Janelle CM. Emotion and movement: activation of defensive circuitry alters the magnitude of a sustained muscle contraction. Neurosci Lett. 2006 Apr 3;396(3):192-6. doi: 10.1016/j.neulet.2005.11.048. Epub 2005 Dec 20. PMID 16376016
- [Background] Moran TP. Anxiety and working memory capacity: A meta-analysis and narrative review. Psychol Bull. 2016 Aug;142(8):831-864. doi: 10.1037/bul0000051. Epub 2016 Mar 10. PMID 26963369
- [Background] Doumas M, Morsanyi K, Young WR. Cognitively and socially induced stress affects postural control. Exp Brain Res. 2018 Jan;236(1):305-314. doi: 10.1007/s00221-017-5128-8. Epub 2017 Nov 14. PMID 29138872
- [Background] MacIntyre TE, Madan CR, Moran AP, Collet C, Guillot A. Motor imagery, performance and motor rehabilitation. Prog Brain Res. 2018;240:141-159. doi: 10.1016/bs.pbr.2018.09.010. Epub 2018 Oct 24. PMID 30390828
- [Background] Schuster C, Hilfiker R, Amft O, Scheidhauer A, Andrews B, Butler J, Kischka U, Ettlin T. Best practice for motor imagery: a systematic literature review on motor imagery training elements in five different disciplines. BMC Med. 2011 Jun 17;9:75. doi: 10.1186/1741-7015-9-75. PMID 21682867
- [Background] Trapero-Asenjo S, Gallego-Izquierdo T, Pecos-Martin D, Nunez-Nagy S. Translation, cultural adaptation, and validation of the Spanish version of the Movement Imagery Questionnaire-3 (MIQ-3). Musculoskelet Sci Pract. 2021 Feb;51:102313. doi: 10.1016/j.msksp.2020.102313. Epub 2020 Dec 9. PMID 33310512
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Derived] Trapero-Asenjo S, Fernandez-Guinea S, Guillot A, Pecos-Martin D, Nunez-Nagy S. Muscle relaxation enhances motor imagery capacity in people with anxiety: A randomized clinical trial. PLoS One. 2025 Jan 10;20(1):e0316723. doi: 10.1371/journal.pone.0316723. eCollection 2025. PMID 39792894